CLINICAL TRIAL: NCT03072264
Title: Randomized Clinical Trial Comparing Mindfulness, Pharmacological Treatment, and Control Group in Generalized Anxiety Disorder (GAD)
Brief Title: Randomized Clinical Trial of a Mindfulness Based Intervention in Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160301
Record Dates: First submitted 2017-01-05; First posted 2017-03-07 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder, GAD, mindfulness, anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Fluoxetine; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Body in Mind Training (BMT) (Experimental): This is a group intervention (10-15 participants) that consists of 5 weekly sessions lasting 2 hours. In our protocol, we added 3 more final sessions of 2 hours in order to emphasize the practices, specially in self-compassion, resulting in 8 weeks of intervention.
  Interventions: Behavioral: Body in Mind Training (BMT)
- Medication (Active Comparator): In this group, individuals will consult with a psychiatrist weekly and will receive fluoxetine in a dosage of 20 to 60mg/dia according to clinical response.
  Interventions: Drug: Fluoxetine
- Quality of Life Group (Active Comparator): This is a group intervention (10-15 participants) that consists of 8 weekly sessions lasting 2 hour in which individuals will receive psychoeducation on various aspects of quality of life that have na impact in reducing anxiety.
  Interventions: Behavioral: Quality of Life Group

INTERVENTIONS:
Behavioral: Body in Mind Training (BMT) — Session 1 - Stop; Session 2 - Intention; Session 3 - Attention; Session 4 - Scientist Myself; Session 5 - Self-Compassion; Sessions 6, 7, 8 - Practice.
  Other Names: Mindfulness Based Intervention
  Arms: Body in Mind Training (BMT)
Drug: Fluoxetine — In this group, individuals will consult with a psychiatrist weekly and will receive fluoxetine in a dosage of 20 to 60mg/dia according to clinical response.
  Other Names: Control Group
  Arms: Medication
Behavioral: Quality of Life Group — Session 1 - Psychoeducation; Session 2 - Substance Use; Session 3 - Sleep; Session 4 - Physical Exercise; Session 5 - Healthy Eating; Sessions 6, 7,8 - discussions.
  Other Names: Control Group
  Arms: Quality of Life Group

SUMMARY:
The literature suggests that Mindfulness Based Intervention may be effective in the treatment of anxiety symptoms. The objective of this study is to compare the clinical effectiveness of a Mindfulness Based Intervention - the Mind in Body Training (MBT) - with a selective serotonin reuptake inhibitor (Fluoxetine) and an active control group (Quality of Life) through different biological and clinical outcomes, as well as evaluate some possible mechanisms of treatment response. Methods: it is a three armed randomized, controlled clinical trial. Participants with General Anxiety Disorder will be recruited. A community sample of 192 participants will be randomly allocated to the MBT, Fluoxetine or Quality of Life Group. Instruments measuring anxiety, worry and meta-worry symptoms, quality of life, acceptance and self-compassion, mindfulness, rumination and emotion regulation will be applied. The patients will be submitted to Error Related Negativity (ERN) and Heart Rate Variability (HRV) measures. The primary outcome is the effectiveness of MBT compared with Fluoxetine and Quality of Life Group in symptomatic outcomes. The secondary outcome are the effectiveness os these interventions in emotional regulation process and biological measures (ERN and HRV), and the evaluation of BMT mechanisms through possible mediation of treatment response for emotional processes like mindfulness, acceptance and self-compassion, biological changes (ERN and HRV), and metacognition.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is the most prevalent Anxiety Disorder after Specific Phobia. It is characterized by persistent and excessive anxiety and worry about different domains of life that is difficult to control, and the individuals can experience physical symptoms, like restlessness or feeling keyed up or on edge, being easily fatigued, difficulty concentrating or mind going blank, irritability, muscle tension, and sleep disturbance. Also, GAD is one of the most common mental disorders in primary care settings, and it is associated with increased use of health care resources and disability, functional impairment, psychiatric and medical comorbidities.

Despite its prevalence and impairment, this disorder is under-recognized, and less than one-third of patients are adequately treated. The literature demonstrates that either psychotropic medications or cognitive behavior therapy (CBT) appear to be effective for treating GAD. However, a substantial number of patients do not respond to initial treatment, and, although the response rates are inconsistent across studies, only 38% of the treated patients have a remission after five years. Moreover, GAD is usually a chronic disorder with a waxing and waning course, requiring a long-term treatment.

In relation to some biological mechanisms in GAD, some studies report an enhanced Error-Related Negativity (ERN) and a lower Heart Rate Variability (HRV) in GAD patients. The first biological marker could be associated with anxious apprehension and the main findings are found in GAD while the second one reflects a reduction in parasympathetic modulation. On the other hand, it is already known that mindfulness meditation practice is associated with increase in autonomic regulation by stimulating the parasympathetic system. In relation to cognitive factors, the literature demonstrates that GAD patients have a higher level of experiential avoidance and distress about emotions, more negative believes about worry and meta-worry.

Mindfulness is a practice developed to foster self-regulation. Historically, the mindfulness exercises used in clinical protocols are linked with the Buddhist framework in which it is a means to alleviate suffering and cultivate compassion. In the West, the role of mindfulness in health promotion has been the target of studies since the 70s and it has been incorporated in cognitive-behavioural treatments. The Body in mind training (BMT) is a treatment protocol that focuses on movement and motor system as a tool for mindfulness practice. More than three decades of studies have shown the positive effects of mindfulness based interventions (MBIs) in both mental and physical health and quality of life either in general population or clinical populations. Also, MBIs seem to be effective and a lasting alternative to treat anxiety. In relation to GAD, some studies have shown that MBI's are effective, but, in generally, they are limited by the small sample size or the use of waiting list control instead of an active control group.

So, the objective of this research is to evaluate the effectiveness of BMT intervention and compared to Fluoxetine and a Quality of Life Group in the treatment of GAD patients. Also, we intend to evaluate some biological and cognitive mechanisms of these different treatments through mediators analysis.

It is a single blind Randomized Controlled Trial with three arms of treatments. The individuals will be recruited in the community. Generalized Anxiety patients (according to Mini-International Neuropsychiatric Interview) will be randomly allocated (in a 1:1:1 ratio) to receive either antidepressant: BMT: Control Group. Research assessors will be masked. Because of the nature of the interventions, patients and clinicians will be aware of treatment allocation. The duration of the treatments is 8 weeks.

Before, in the week 5, and after the interventions, participants will be assessed with the Hamilton Anxiety Rating Scale (HAM-A), Clinical Global Impression (CGI), Anxiety Sensitivity Index (ASI), Penn State Worry Questionnaire (PSWQ), Difficulties in Emotion Regulation Scale (DERS), Five Facet Mindfulness Questionnaire (FFMQ), Self-Compassion Scale (SCS), Action and Acceptance Questionnaire (AAQ), Ruminative Response Scale (RRS), Metacognition Questionnaire (MCQ-30), Meta-worry Questionnaire (MWQ), WHOQOL-Bref. Also, before the interventions, participants will answer the Early Life Experiences Scale (ELES) and Early Memories of Warmth and Safeness Scale (EMWSS). The HRV and ERN will be assessed before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old;
* Primary Generalized Anxiety Disorder (GAD) according to M.I.N.I;
* Possibility to attend the Hospital every week during 8 weeks.

Exclusion Criteria:

* Current psychopharmacological or psychotherapeutic treatment for GAD;
* Previous no response treatment with fluoxetine for GAD;
* Bipolar Disorder, Psychotic Disorder, Substance Use Disorder (except tobacco) in the last 6 months or Suicidal Ideation in the last 6 months (M.I.N.I);
* Hamilton Depression Scale (HAM-D) ≥23;
* Any contraindication to fluoxetine use;
* Clinical instability or immobility;
* Pregnancy or lactation;
* Antisocial Personality Disorder;
* Eating Disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline in Penn State Worry Questionnaire (PSWQ) Score | Baseline , 8 weeks
  Efficacy Assessment
Mean Change From Baseline in Hamilton Anxiety Scale (HAM-A) Score | Baseline , 8 weeks
  Efficacy Assessment

SECONDARY OUTCOMES:
Mean Change From Baseline in Heart Rate variability (HRV) | Baseline , 8 weeks
  Biological Efficacy Assessment 1
Mean Change From Baseline in Error-Related Negativity (ERN) | Baseline , 8 weeks
  Biological Efficacy Assessment 2
Mean Change From Baseline in Quality of Life (WHOQOL) Scores | Baseline , 8 weeks
  Efficacy Assessment in Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Gisele Gus Manfro, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costa MA, Goncalves FG, Tatton-Ramos T, Fonseca NKOD, Schwinn JK, Alves SG, Salum GA, Manfro GG. A Three-Arm Randomized Clinical Trial Comparing the Efficacy of a Mindfulness-Based Intervention with an Active Comparison Group and Fluoxetine Treatment for Adults with Generalized Anxiety Disorder. Psychother Psychosom. 2021;90(4):269-279. doi: 10.1159/000511880. Epub 2020 Dec 15. PMID 33321509